CLINICAL TRIAL: NCT04014946
Title: Prospective Assessment of Risk Factors for Appropriate ICD Intervention in Patients With Ischemic Cardiomyopathy
Brief Title: Assessment of Risk Factors for Appropriate ICD (Implantable Cardioverter-defibrillator) Intervention in Patients With Ischemic Cardiomyopathy
Acronym: PARCADIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TA97
Record Dates: First submitted 2019-05-10; First posted 2019-07-10 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: ICD; Cardiomyopathy Ischemic; Primary Prevention

STUDY DESIGN:
Intervention Model Description: The study model is single group. At the analysis the patients will be divided in two groups bij outcome of ICD therapy/no ICD therapy.
  The endpoints related to the primary hypothesis are appropriate ICD intervention (shock or ATP) and Relative Infarct Transmurality (RIT = transmural infarct mass / total infarct mass) obtained from LGE-CMR. ICD interventions will be labeled appropriate or non-appropriate by an independent endpoint committee.
  * RITshock or ATP: RIT expectation value in patients with ≥1 appropriate shock or ATP therapy until the 24mo follow-up
  * RIT no shock or ATP: RIT expectation value in patients without any appropriate shock or ATP therapy until the 24mo follow-up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICD implantation (Other): Implantation of a Lumax 540 single/dual chamber ICD or successor according to local practice within 3 months after enrolment. The patient will be implanted with a single or dual chamber device according to ESC guidelines.
  Interventions: Device: ICD implantation

INTERVENTIONS:
Device: ICD implantation — implantation of the Lumax 540 single/dual chamber ICD or successor
  Other Names: Lumax 540 single/dual chamber ICD or successor

SUMMARY:
Design: PARCADIA is a prospective non-randomized non-interventional multi-center clinical investigation in Europe. Patients with depressed LV (left ventricular) function assessed on local standards, of ischemic origin and on chronic optimal medical therapy will be selected according to inclusion and exclusion criteria, implanted with an ICD after executing baseline investigations and prospectively followed up for minimal 24 months and until the termination of the clinical investigation.

General objective: analysis of baseline risk factors to identify predictors for appropriate ICD intervention in patients with ischemic cardiomyopathy receiving an ICD for primary prevention (MADIT II population).

Hypothesis: The primary alternative hypothesis states that the mean relative infarct transmurality (RIT) is different in patients with (RITshock or ATP (Anti Tachy Pacing)) and without (RITno shock or ATP )appropriate ICD intervention, i.e. shock or ATP.

* Null hypothesis (H0): RITshock or ATP = RITno shock or ATP
* Alternative hypothesis (Ha): RITshock or ATP ≠ RITno shock or ATP

Sample size: 200 patients.

Follow-up: Enrolment visit, pre implant screening, ICD implantation, pre-hospital discharge visit, and follow-up (FUP) visits at 2, 6, 12, 18, 24 months including home monitoring. Additional routine FUP every 6 months until study termination after last enrolled patient has completed 2 years FUP.

DETAILED DESCRIPTION:
Rationale: Implantation of an ICD as primary prevention therapy is indicated according to the current guidelines based on the low LVEF (Left Ventricular Ejection Fraction) as it was shown to significantly reduce mortality. Although of proven efficacy, ICD therapy is associated with survival benefit in only a small fraction of patients. It is estimated that 18 patients would have to receive an ICD to save one life, resulting in a huge burden on national health systems. Moreover, only about one quarter of all guideline eligible primary prevention ICD patients receive appropriate shocks. The above considerations support the need for an effective risk-stratification method to identify patients that benefit most (or least) from this therapy. Evaluation of ventricular anatomy and function by imaging techniques has become more important since this provides information on the substrate (myocardial scar) and trigger of life-threatening ventricular arrhythmias. Besides accurate estimation of left and right ventricular volumes and functions, Late Gadolinium Enhanced Cardiac Magnetic Resonance (LGE-CMR) imaging has a very high sensitivity to detect myocardial scar. Quantification of scar characteristics by cardiac MRI might be useful for the prediction of future arrhythmic events in patients with ischemic cardiomyopathy. However evidence is conflicting and published papers are hampered by limited patient numbers and can only be regarded in the light of generating hypothesis. The PARCADIA clinical investigation will explore the potential of cardiac MRI as a predictor for appropriate ICD intervention in a multicenter setting.

PARCADIA is a prospective non-randomized non-interventional multi-center clinical investigation in Europe. Patients with depressed LV (Left Ventricular) function assessed on local standards, of ischemic (at least 40 days post-MI (myocardial infarction) or 3 months post revascularization) origin and on chronic optimal medical therapy will be selected according to inclusion and exclusion criteria, implanted with an ICD after executing baseline investigations and prospectively followed up for minimal 24 months and until the termination of the clinical investigation

General objective: analysis of baseline risk factors to identify predictors for appropriate ICD intervention in patients with ischemic cardiomyopathy receiving an ICD for primary prevention (MADIT II population).

The primary objective of the clinical investigation is to determine whether there is a relationship between appropriate ICD intervention (shock or ATP) and the Relative Infarct Transmurality (RIT) obtained from Late Gadolinium Enhanced Cardiac Magnetic Resonance (LGE-CMR) imaging in patients with ischemic cardiomyopathy, receiving an ICD for primary prevention.

Methodology: Screening: (within 6 months before enrolment) patients with LV depressed function due to Ischemic Cardiomyopathy with an indication for primary prevention ICD implantation according to ESC (European Society of Cardiology) guidelines or local standards will be screened within 6 months before enrolment.

pre implant diagnostics: within 3 months after enrolment LGE-CMR imaging, 24h holter, 12-lead ECG, will be performed and biochemical markers will be obtained.

ICD implantation: Implantation of a Lumax 540 single/dual chamber ICD or successor withiin 3 months after enrolment. The ICD will be programmed according to protocol.

Pre-hospital discharge an ICD interrogation wil be performed. Follow-up (FUP) visits at: 2, 6, 12, 18, 24 months with inclusion of standard 12-lead ECG, ICD check-up and cardiologist visit in the outpatient clinic. Additional routine FUP every 6 months until study termination after last enrolled patient has completed 2 years FUP.

ELIGIBILITY:
Inclusion Criteria:

* Patient with ischemic cardiomyopathy indicated for a de novo ICD implantation for primary prevention, according to ESC guidelines or local standards (MADIT II population)
* Written informed consent / willingness and ability to comply with the protocol

Exclusion Criteria:

* Contraindication for MRI
* Severe renal dysfunction (stage 4 or 5) resulting in contra-indication for the admission of gadolinium during MRI (See Appendix A for more details)
* Indication for secondary prevention ICD implantation
* Class I indication for cardiac resynchronization therapy
* Heart failure with New York Heart Association functional class IV
* LV ejection fraction >40%
* Age <18 years and >85 years
* Women that are pregnant, lactating or planning to become pregnant
* Participating in any other clinical trial with active intervention(s) during the course of this study
* Life expectancy less than 1 year

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-07-22 (Actual)

PRIMARY OUTCOMES:
Relative Infarct Transmurality | Measured during Late gadolinium enhancement cardiovascular magnetic resonance (LGE-CMR) imaging within 3 months after inclusion and before ICD implantation
  Percentage Relative Infarct Transmurality (RIT = transmural infarct mass / total infarct mass) obtained from LGE-CMR
appropriate ICD intervention (shock or ATP) | Until the 24 month follow-up
  assessment whether patient had appropriate ICD intervention (shock or ATP) or not during 24 months follow-up. ICD interventions will be labeled appropriate or non-appropriate by an independent endpoint committee.

SECONDARY OUTCOMES:
LV function (EF) | Baseline
  Left Ventricular function (Ejection Fraction in %) measured during LGE-CMR at baseline before ICD implantation
LV mass | Baseline
  LV mass measured during LGE-CMR at baseline before ICD implantation
total infarct mass | Baseline
  total infarct mass measured during GGE-CMR at baseline before ICD implantation
transmural infarct mass | Baseline
  transmural infarct mass measured during LGE-CMR at baseline before ICD implantation
mean Heart Rate (HR) | Baseline
  mean HR measured by 24-hrs Holter
Day and night HR | baseline
  Day and night HR measured by 24-hrs Holter
spontaneous episodes of atrial and ventricular arrhythmias | baseline
  number of spontaneous episodes of atrial and ventricular arrhythmias measured by 24-hrs Holter
heart rate variability (SDNN: Standard deviation of consecutive normal-to-normal intervals) | baseline
  heart rate variability (SDNN) measured by 24-hrs Holter
HR | baseline
  HR on 12 lead ECG
rhythm | baseline
  rhythm on 12 lead ECG
QRS width | baseline
  QRS width on 12 lead ECG
serum sodium and potassium | baseline
  concentration of serum sodium and potassium (in mmol/l ) (blood sample)
serum creatinine | baseline
  concentration of serum creatinine (in umol/l) (blood sample)
uric acid | baseline
  concentration of uric acid (in mmol/l) (blood sample)
albumin | baseline
  concentration of albumin (in g/l) (blood sample)
HbA1c (Hemoglobin A1c) | baseline
  concentration HbA1c (mmol/mol) (blood sample)
NT-proBNP (N-terminal pro-hormone Brain Natriuretic Peptide) | baseline
  concentration NT-proBNP (in pg/ml) (blood sample)
hsTNT/I (high sensitive Troponin-T/I) | baseline
  concentration hsTNT/I (in ng/ml) (blood sample)
aldosterone | baseline
  concentration aldosterone (in pmol/l) (blood sample)
incidence of hypertension | baseline
  Baseline clinical demographics: hypertension in clinical history
incidence of diabetes | baseline
  Baseline clinical demographics: diabetes in clinical history
incidence of hypercholesterolemia | baseline
  Baseline clinical demographics: hypercholesterolemia in clinical history
PVC/hr: Premature ventricular contraction per hour | baseline
  PVC/hr: Premature ventricular contraction per hour on 24hrs Holter

IPD SHARING:
Plan to Share IPD: No